CLINICAL TRIAL: NCT06688331
Title: A Multicenter, Randomized, Blinded, Placebo Controlled, Phase II Study to Evaluate the Safety and Efficacy of Cell Therapy Based With Artificially Expanded CD4+CD25+CD127- Regulatory Lymphocytes and Anti-CD20 Antibody in Pediatric Patients With Presymptomatic Diabetes Type 1 (Stage 1)
Brief Title: Treatment of Presymptomatic (Stage 1) Type 1 Diabetes Pediatric Patients With Treg Cell Preparations and Anti-CD20 Antibody
Acronym: PreTreg
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PolTREG S.A. (Industry)
Collaborators: Invicta Sp. z o.o. (Other); Medical Research Agency, Poland (Other Government); Clinmark Clinical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PTG007-DM1-preTREG-001; 2023-505226-33-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Presymptomatic Diabetes Type 1 (Stage 1); Diabetes Mellitus, Type I; Diabetes Mellitus, Type 1
Keywords: PreTreg; Tregs; Prediabetes; presymptomatic
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Prediabetic State | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: Trial type: Prospective randomized, placebo-controlled, parallel group, blinded trial.
  Control method: placebo, active comparator, sham procedure.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding: The following roles indicated below will not be made aware of the treatment group assignment during the trial:
  * participant
  * legal representatives
  * site staff excluding pharmacists (applies to anti-CD20 only)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TregsCD20 (Experimental): Infusion of Treg preparation at "day 0" + 4 doses of antiCD20 antibody; second infusion of Treg preparation at time "+90±30days" Interventions: ex vivo expanded CD4+CD25+CD127- regulatory T cells (Tregs) + Anti-CD20 (rituximab)
- Tregs only (Experimental): Infusion of Treg preparation at "day 0" + 4 doses of placebo; second infusion of Treg preparation at time "+90±30 days"
  Interventions: Biological: ex vivo expanded CD4+CD25+CD127- regulatory T cells (Tregs); Other: Placebo
- CD20 only (Experimental): Infusion of Treg sham at "day 0" + 4 doses of antiCD20 antibody; second infusion of Treg sham at time "+90±30days"
  Interventions: Biological: Anti-CD20 (rituximab); Other: Treg sham
- Control group (Placebo Comparator): Infusion of Treg sham at "day 0" + 4 doses of placebo; second infusion of Treg sham at time "+90±30days"
  Interventions: Other: Placebo; Other: Treg sham

INTERVENTIONS:
Biological: ex vivo expanded CD4+CD25+CD127- regulatory T cells (Tregs) — regulatory T cells with the phenotype CD3(+)CD4(+)CD25(high)CD127(-)doublet(-)lin(-)
  Other Names: Tregs; regulatory T cells
  Arms: Tregs only
Biological: Anti-CD20 (rituximab) — rituximab
  Other Names: Mabthera
  Arms: CD20 only
Other: Placebo — intrevenous 0,9% NaCl
  Arms: Control group; Tregs only
Other: Treg sham — intrevenous 0,9% NaCl
  Arms: CD20 only; Control group

SUMMARY:
The main purpose of the study is to check:

* Can therapy with a preparation of regulatory cells (Tregs lymphocytes) and/or an anti-CD20 antibody preparation (rituximab) be successfully used in children with pre-diabetes to treat or delay type 1 diabetes?
* Is therapy with a preparation of regulatory cells (Tregs lymphocytes) and/or a preparation of antiCD20 antibodies (rituximab) safe for children with pre-diabetes, and what side effects may be associated with it? The study will include patients at high risk for type 1 diabetes whose laboratory tests have confirmed preserved normal/high insulin production. First (part 1 of the study), tests will be performed to determine the risk of the disease (determination of autoantibodies that characterize the autoimmune background).

In order to confirm the effectiveness of the therapy, not all patients will receive the study treatment. The study will be a so-called blinded randomized trial. This means that in this trial, all participants will undergo the same study procedures, but the participant will be randomly assigned to one of four (4) groups that will receive different treatment regimens before entering the study.

The participant will be randomly assigned to one of four groups:

* Group I will receive a preparation of regulatory cells (Tregs lymphocytes) along with a preparation of antiCD20 antibodies,
* Group II will receive a preparation of regulatory cells (Tregs lymphocytes) together with an inert substance (placebo)
* Group III will receive a preparation of antiCD20 antibodies along with a sham treatment (inert substance)
* Group IV will receive an agent containing an inert substance and sham treatment.

Approximately 150 patients aged 6-16 who are at risk of developing type 1 diabetes will be enrolled in the study, which will last up to 96 months. Each enrolled participant will remain in the study for up to five years.

DETAILED DESCRIPTION:
Participants: screening of approximately 2500 high-risk subjects will be conducted until no less than 150 participants with confirmed stage 1 (preclinical) type 1 diabetes mellitus are randomized; randomization 2:1:1:2; 50 participants treated with Tregs and anti-CD20 antibody; 25 participants treated with Tregs; 25 participants treated with anti-CD20 antibody; control: 50 participants receiving placebo and sham Tregs.

Inclusion of participants: up to 36 months. Trial intervention: Total duration of the trial intervention for each participant will be approximately 3 Months. After completion of the trial intervention, participants will be monitored at the sites for the onset of type 1 diabetes mellitus for a maximum of five years counting from the first dose of Tregs.

Follow-up time: post-treatment observation of all participants to 57 months (day "0" is the day of administration of the first dose of Treg/sham preparation).

Trial time: 96 months. Trial type: Prospective randomized (phase 2), placebo-controlled, parallel group, blinded trial.

Blinding: The following roles indicated below will not be made aware of the treatment group assignment during the trial:

* participant
* legal representatives
* site staff excluding pharmacists (applies to anti-CD20only)

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-16
2. 25 ≤ BMI ≤ 75 percentile (acc. to OLAF) with a lower weight threshold of 20 kg
3. Venous plasma glucose levels < 100mg% at fasting (70 to 100 mg/dl) and normal glucose tolerance test (at 120 minutes glycaemia <140 mg/dl) (acc. to PTD)
4. Insulin independence
5. C-peptide levels ≥ 1.0 ng/ml (central laboratory limit of normal) in fasting and post-stimulation tests increase ≥ 100%
6. Participant has not yet been diagnosed with stage 2 or 3 type 1 diabetes mellitus (no history of dysglycemia, no history of clinical symptoms of type 1 diabetes mellitus)
7. HbA1c level (%) <5,7% (acc. to ADA)
8. Positive autoantibody titres (ICA, IAA, GAD, IA-2/ICA512, ZnT8) - low titers of two or more antibodies (2-4 times the normal*); if high titer of one of the antibodies (≥ 4 times the norm, not applicable to ICA) re-screening allowed (the participant can be included in the trial only after confirming two or more antibodies)
9. Ability to give informed consent by the child's legal representatives (and the child himself or herself if he or she is over the age of 13 at the time of the trial [according to local law])
10. Ability of the child's legal representatives to manage diabetes, defined as blood glucose levels control at least three times a day and the ability to dose insulin correctly.
11. Venous access to guarantee blood donation

    Exclusion Criteria:
12. Refusal to participate in the trial or lack of a signed informed consent form
13. Suspicion or diagnosis for a type of diabetes other than type 1 diabetes mellitus
14. Age under 6 or above 16
15. IgA deficiency or history of other diagnosed immunodeficiency (max. 7 infections/year allowed, and the prognosis should indicate that the patient will remain in the study throughout its duration)
16. C-peptide levels < 1.0 ng/ml fasting and in post-stimulation tests increase < 100%
17. Glucose levels in venous blood ≥ 100mg% fasting
18. Glucose levels in venous blood after 1 and 2 hours in OGTT ≥ 200mg%
19. Glycated hemoglobin level (HbA1c) in venous blood ≥ 5,7%
20. BMI < 25 or > 75th percentile for a given age or weight of less than 20 kg
21. History of hypersensitivity to anti-CD20 or other components of the preparation
22. History of hypersensitivity to penicillin and/or streptomycin
23. Past or active infection with HBV, HCV, HIV, HTLV I/II, mycobacterium tuberculosis, syphilis. Laboratory evidence of infection without the need for clinical signs and symptoms is sufficient for diagnosis.
24. Active infection with the EBV or CMV virus (positive IgM)
25. Any fungal, parasitic, viral, or bacterial infection
26. History of past or active cancer
27. Anemia, lymphopenia, neutropenia, or thrombocytopenia defined as a blood cell count below the lower limit of normal for age found within the last 6 weeks prior to trial inclusion
28. Elevated thrombotic activity/history of thrombosis episode
29. Any disease prior to inclusion in the trial currently requiring medication for more than 3 months in history
30. Diagnosed autoimmune disease other than type 1 diabetes mellitus, including a history of Hashimoto's disease and coeliac disease
31. Taking anti-diabetic medication (including insulin) in the last 4 weeks prior to trial inclusion
32. History of retinopathy
33. History of hypertension
34. Current or history of albuminuria
35. For women in childbearing potential/menstruating women: pregnancy (from medical interview) or unwillingness to exercise sexual restraint or use effective forms of contraception for the duration of the trial and up to 4 months after completion, if applicable.

    The following contraceptive methods are acceptable: bilateral fallopian tube closure, sterilization in men, appropriate use of hormonal contraception that inhibits ovulation, hormone-releasing IUDs, and copper IUDs, male or female condoms with spermicide; and cap, uterine disc, or sponge with spermicide.
36. Breastfeeding
37. For males over 15 years of age: expressed intention to have offspring or donate sperm during the trial or within 4 months after the end of the trial, if applicable
38. Excessive anxiety of the participant or his/her legal representatives regarding the procedures used in the trial
39. Any medical problem that, in the opinion of the investigator, may adversely affect the participant's health if included in the trial
40. Legal representatives and/or children over the age of 15 with an identified alcohol and/or psychoactive substance addiction
41. History of disease of unknown etiology
42. History of Creutzfeldt-Jacob disease
43. History of progressive dementia or degenerative neurological disease, including of unknown origin
44. History of taking hormones derived from the human pituitary gland (e.g., growth hormone)
45. Treatment with immunosuppressants
46. History of corneal, scleral, and dural transplant or undocumented neurosurgery
47. History of occurrence of risk factors related to the participant's travel, where there is a possibility of exposure to regional infectious diseases
48. Physical signs that indicate the risk of an infectious disease
49. History of xenogeneic transplant

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Number of days from day 0 to the day of first dysglycemia (stage 2 of type 1 diabetes mellitus) in each group | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  To assess the safety and efficacy of the treatment used in the separate groups of participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/Tregs sham)
Number of adverse events reported 1 year, 2 years after the first dose of Tregs and at the end of the trial | From enrollment to the end of participation in the trial at month 60 (day "0" is the day of administration of the first dose of Treg preparation)
  To assess the safety and efficacy of the treatment used in the separate groups of participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/Tregs sham)

SECONDARY OUTCOMES:
Percentage of participants in each group who are in stage 2 type 1 diabetes mellitus, i.e., presence of autoantibodies, dysglycemia or stage 3 at year 1 and every year thereafter after the first dose of Tregs/placebo | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  Additional measures to assess the safety and efficacy of the treatment used in the separate groups of pediatric participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/ Tregs sham) in preserving β-cell function
Total number of days from the date of diagnosis of stage 2 to the date of onset of full-blown type 1 diabetes mellitus (stage 3 of type 1 diabetes mellitus) in each group (normalized to the number of person/days in each group) | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  Additional measures to assess the safety and efficacy of the treatment used in the separate groups of pediatric participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/ Tregs sham) in preserving β-cell function
C-peptide levels [fasting/post MMTT stimulation (AUC) 1 year, 2 years after the first dose of Tregs and then annually until the end of the trial | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  Additional measures to assess the safety and efficacy of the treatment used in the separate groups of pediatric participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/ Tregs sham) in preserving β-cell function
Daily dose of insulin per kg body weight (DDI) 1 year, 2 years after the first dose of Tregs, and annually thereafter until the end of the trial | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  Additional measures to assess the safety and efficacy of the treatment used in the separate groups of pediatric participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/ Tregs sham) in preserving β-cell function
Number of participants in remission 1 year, 2 years after the first dose of Tregs, and annually thereafter until the end of the trial, [remission defined as daily insulin dose is less than 0.5U/kg/day with an HbA1c level less than 6.5%] | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  Additional measures to assess the safety and efficacy of the treatment used in the separate groups of pediatric participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/ Tregs sham) in preserving β-cell function
Assessment of the incidence and severity of adverse events associated with the administration of Treg preparation or antiCD20 antibody, primarily the effects of immunosuppression: incidence of infections of any etiology and de novo tumors detected | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  Additional measures to assess the safety and efficacy of the treatment used in the separate groups of pediatric participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/ Tregs sham) in preserving β-cell function
Percentage of participants in each group who are still in stage 1 type 1 diabetes mellitus, i.e., presence of autoantibodies and normoglycemia | From day "0" (the day of administration of the first dose of Treg preparation) to the end of participation in the trial at month 60
  Additional measures to assess the safety and efficacy of the treatment used in the separate groups of pediatric participants treated with combined treatment with Treg preparation and rituximab antibody or Treg preparation or rituximab antibody or the control (placebo/ Tregs sham) in preserving β-cell function

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Trzonkowski, Prof, Study Director — PolTREG S.A.; Artur Bossowski, Prof, Principal Investigator — Uniwersytecki Dzieciecy Szpital Kliniczny Im. L. Zamenhofa W Bialymstoku; Wojciech Mlynarski, Prof, Study Chair — Uniwersytet Medyczny W Lodzi
Locations (8):
- Poland (8):
  - Uniwersytecki Dzieciecy Szpital Kliniczny Im. L. Zamenhofa W Bialymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Gornoslaskie Centrum Zdrowia Dziecka Im. Sw. Jana Pawla II Samodzielny Publiczny Szpital Kliniczny Nr 6 Slaskiego Uniwersytetu Medycznego W Katowicach, Katowice
  - Uniwersytet Medyczny W Lodzi, Lodz
  - Uniwersytecki Szpital Dzieciecy w Lublinie, Lublin
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - Centrum Medyczne Medyk Sp. z o.o. S.K., Rzeszów
  - Uniwersytecki Szpital Kliniczny Im. Jana Mikulicza-Radeckiego We Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CTIS — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-505226-33-00